CLINICAL TRIAL: NCT06211998
Title: Comparison of Mesh Nebulizer and Compressor Nebulizer on Pulmonary Function Test in Children Presenting With Asthma Attack: A Double-Blind Randomized Comparative Clinical Trial
Brief Title: Comparison of Mesh Nebulizer and Compressor Nebulizer With Pulmonary Function Test in Pediatric Asthma Attacks
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Berker Okay (Other)
Responsible Party: Sponsor-Investigator, Berker Okay, M.D., Haseki Training and Research Hospital
Organization: Haseki Training and Research Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 140-2022
Record Dates: First submitted 2023-12-25; First posted 2024-01-18 (Actual); Last update posted 2024-01-18 (Actual); Status verified 2024-01

CONDITIONS: Asthma; Asthma in Children
Keywords: Asthma; Child; Compressor Nebulizer; Mesh Nebulizer; Pulmonary function test
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group receiving inhaled treatment with compressor nebulizer (Active Comparator): Salbutamol inhaler, Omron® CompAIR Pro NE-C900 Compressor Nebulizer (Omron Healthcare Co., Ltd., Kyoto, Japan) was used in Group 1
  Interventions: Device: Group 1
- Group receiving inhaled treatment with mesh nebulizer (Active Comparator): Salbutamol inhaler, Mesh nebulizer (Aerogen Solo®, Aerogen Ltd, Galway, Ireland) was used in Group 2
  Interventions: Device: Group 2

INTERVENTIONS:
Device: Group 1 — Salbutamol inhaler, Omron® CompAIR Pro NE-C900 Compressor Nebulizer (Omron Healthcare Co., Ltd., Kyoto, Japan) was used in Group 1
  Arms: Group receiving inhaled treatment with compressor nebulizer
Device: Group 2 — Salbutamol inhaler, Mesh nebulizer (Aerogen Solo®, Aerogen Ltd, Galway, Ireland) was used in Group 2
  Arms: Group receiving inhaled treatment with mesh nebulizer

SUMMARY:
Asthma is a worldwide health problem and is one of the most common chronic diseases of childhood in most countries. Symptoms begin before the age of 5 years in 80% of children with asthma, but the diagnosis is not always easy. The National Asthma Education and Prevention Program (NAEPP) expert panel recommends spirometry testing for children over 5 years of age. Spirometry measurements include forced vital capacity (FVC) and the forced expiratory volume in first second (FEV1). Airflow obstruction is defined as FEV1 reduced to less than 80 percent predicted and an FEV1/FVC ratio of less than 0.85 (85 percent). Reference values are based on age, height, sex, and race. Forced expiratory flow between 25 and 75 percent of vital capacity (FEF25-75) less than 65 percent correlates with reversible airflow obstruction in children with normal FEV1 and may be a useful measure in this subgroup.

In the spirometry test, FEV1, FVC, FEF 25-75% values are valuable for the follow-up of asthma. While the FEV1/FVC ratio is above 80% in healthy children, it may decrease below 75% in diseases such as asthma. Likewise, FEV1 and FEF can be found to be low in 50-75% of asthma patients. In addition, these values can be used to determine the effectiveness of the inhaler given with the nebulizer given during the attack. Spirometry should be performed before and after administration of a bronchodilator to assess for reversibility (bronchodilator response [BDR]) even in children with a normal baseline FEV1 because many of these children will still have a BDR (both within the normal range and sometimes also supranormal) after treatment. Significant reversibility is indicated by an increase in FEV1 of ≥12 percent from baseline after administration of a short-acting bronchodilator. This definition for BDR positivity was established primarily in adults. An increase in FEV1 of ≥8 percent may be a better definition for BDR in children.

Inhaled short-acting beta-2 agonists, particularly albuterol (salbutamol), are the standard emergent treatment for acute asthma exacerbations in all patients based upon adult data. It is recommended to be given every 20 minutes in case of need for repeated doses in mild and moderate asthma attacks. Different types of nebulizers can be used for inhaler therapy; they can convert drugs into vapor form with sound waves, compressed air or by using electrical energy. While compressor nebulizers convert the liquid drug into aerosol form with compressed air, mesh nebulizers convert the drug into aerosol form with the vibrations they create with the help of electrical energy. Mesh nebulizers are more effective than other types of nebulizers, and the amount left in the chamber is less than other models, and it can decompose the drug into smaller particles and reach the more extreme branches of the lung.

In our study, the investigators aimed to determine which nebulizer type is more effective by comparing the effects of mesh nebulizer and compressor nebulizer on spirometry test in children presenting with asthma attack. Thus, the investigators planned to find the most comfortable and effective method for patients by determining the appropriate nebulization technique for patients.

ELIGIBILITY:
Inclusion Criteria:

* Asthma attack patients who need inhaler therapy (salbutamol)
* Patients aged 7-15 years and whose families gave consent for the study

Exclusion Criteria:

* Patients with neuromotor impairment
* Patients with underlying chronic disease (neurological disease such as epilepsy or congenital heart disease)
* Patients with obesity or malnutrition (to equalize drug dose efficacy)
* Patients with those receiving adrenaline, budesonide or ipratropium bromide therapy
* Patients who have used a long-acting bronchodilator in the last 12 hours or a short-acting bronchodilator in the last 2 hours
* Patients with fever above 37.5°C
* Patients with a saturation value below 92% at the time of admission
* Patients with severe asthma attack
* Patients with respiratory failure
* Patients who had problems in performing the test (such as mental retardation, patient incompatibility)
* Patients with diseases involving the chest muscles and those with chronic lung diseases (such as cystic fibrosis, bronchiectasis)

Ages: 7 Years to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 80 (Actual)
Dates: Start 2022-08-01 (Actual); Primary Completion 2023-07-15 (Actual); Study Completion 2023-08-01 (Actual)

PRIMARY OUTCOMES:
Mesh nebulizer improves pulmonary function test results more effectively in children | 1 hour
  Pulmonary function test results in children using mesh nebulizers may be improving more effectively.
  To compare mesh and compressor nebulizers, we planned to compare FEV1, FVC, FEV1/FVC, FEF 25-75 and PEF in pulmonary function testing.

CONTACTS AND LOCATIONS:
Locations (1):
- UHS Haseki Training and Research Hospital, Istanbul, Sultangazi, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Dunne RB, Shortt S. Comparison of bronchodilator administration with vibrating mesh nebulizer and standard jet nebulizer in the emergency department. Am J Emerg Med. 2018 Apr;36(4):641-646. doi: 10.1016/j.ajem.2017.10.067. Epub 2017 Oct 31. PMID 29167030
- [Background] Pitance L, Vecellio L, Leal T, Reychler G, Reychler H, Liistro G. Delivery efficacy of a vibrating mesh nebulizer and a jet nebulizer under different configurations. J Aerosol Med Pulm Drug Deliv. 2010 Dec;23(6):389-96. doi: 10.1089/jamp.2010.0816. Epub 2010 Oct 19. PMID 20958144
- [Background] Yuksel H, Yasar A, Acikel A, Topcu I, Yilmaz O. Two different methods of lidocaine inhalation before diagnostic flexible bronchoscopy: effects on post-bronchoscopy respiratory symptoms. Turk J Med Sci. 2021 Aug 30;51(4):2101-2106. doi: 10.3906/sag-2012-130. PMID 34013705
- [Derived] Okay B, Hatipoglu HU, Okay ZU, Sahin K, Yasar A. Comparing mesh and compressor nebulizers in pulmonary function test in pediatric asthma attacks: A double-blind randomized comparative clinical trial. Respir Med. 2025 Mar;238:107966. doi: 10.1016/j.rmed.2025.107966. Epub 2025 Jan 28. PMID 39884589